CLINICAL TRIAL: NCT05959824
Title: Devintec OR-AT0222 Oral Gel for the Treatment of Canker Sores: A Double Blind, Randomized, Placebo Controlled Clinical Investigation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Devintec Sagl (Industry)
Collaborators: Meditrial SrL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNT2022-01
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Recurrent Aphthous Ulcer
Keywords: aphthous ulcer; canker sores; aphthous stomatitis; Topical oral gel
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind, placebo controlled clinical study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Treatment with OR-AT0222
  Interventions: Device: OR-AT0222
- Group 2 (Placebo Comparator): Treatment with Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Device: OR-AT0222 — Topical viscous gel containing tamarind seed polysaccharide and isolated pea proteins will be used 3 times a day away from the main meals (breakfast lunch and dinner) for 7 days.
  Arms: Group 1
Other: Placebo — Topical placebo viscous gel will be used 3 times a day away from the main meals (breakfast lunch and dinner) for 7 days.
  Arms: Group 2

SUMMARY:
Canker sore, also known as aphthous stomatitis or ulcers and aphthae, is a common ailment, idiopathic in nature, with recurrent painful aphthous ulcers on the non-keratinized oral mucous membranes.

Recurrent aphthous ulcer has higher prevalence in young adults and the frequency decreases with increasing age. The etiology of aphthous ulcer remains unclear. Other possible factors include trauma, drug use, deficiency in vitamin B12, folic acid, iron, stress, hormonal changes and metabolic diseases. Topical agents such as local antibiotics, local antiseptics, NSAIDs, and corticosteroids are generally prescribed for symptomatic relief. Several approved drug formulations such as pills, mouthwash, sprays and paste such as vitamin B12, chlorhexidine mouthwash, steroid lozenges and local anesthetics are primarily suggested for the treatment of aphthous ulcer. Despite the available local treatments, still sometimes oral canker sores may represent a painful burden for the patient and the gel OR-AT0222 may represent a topical product easy to use, well tolerated and effective local pain reliever, by facilitating the healing of the lesion(s).

The Sponsor, Devintec Sagl, presents OR-AT0222, indicated for the management of canker sores, aphthous stomatitis and small lesions of the mouth. The gel forms a persistent protective film with a "barrier effect" that promotes wound healing and protects the lesions of the oral cavity from contact with external agents, providing pain relief and reducing the risk of further irritation.

DETAILED DESCRIPTION:
Each subject will be asked to sign the Informed Consent Form (ICF). A total of 46 subjects will be enrolled, 23 for each group will be randomized with a 1:1 ratio and allocated to one treatment group (blinded assignment). Group 1: Treatment with OR-AT0222 and Group 2: Treatment with Placebo. The patients will be asked to apply 1-2 drops of the gel on their ulcers three times a day for 7 days and to record the aphthous pain level based on visual analogue scale (VAS) using a number scale from 0 to 10, with 0 no pain at all and 10 the most severe pain. The patients have to refrain from eating and drinking for at least 30 minutes after gel application. The study will also assess tolerability and safety (adverse events). At day 8, the patients will be examined again. Complete healing (the time when the pseudomembrane and the erythematous border disappear) will be confirmed by clinician examination at the end of the treatment period. Reduction of the number of ulcers respect to baseline and percent of lesions with complete healing will be also assessed

ELIGIBILITY:
Inclusion Criteria:

1. >18 years (male and females)
2. Patients have one oral canker sore, at least. Onset within 48 hours
3. Patients in good condition with no serious systemic disease

Exclusion Criteria:

1. Hypersensitivity to any OR-AT0222 ingredients
2. Use of any medication to treat the ulcers the previous week before ORAT0222 gel use started or use of local medication or systemic drug during the treatment with OR-AT0222 gel.
3. Underlying systemic disease(s) or a history of immunologic disorder(s);
4. Taking immunomodulatory agents or systemic nonsteroidal antiinflammatory drugs < 1 month before study commencement;
5. Smokers;
6. Could not provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
VAS score | 3xday, 30 minutes after each application for 7 days
  Mean daily pain VAS score of the treatment group vs placebo.

SECONDARY OUTCOMES:
Daily pain VAS score | 5, 10, 15 and 30 minutes after the first (morning) application of the gel, from baseline up to day 7
  Daily pain VAS score at different time points
Pain disappearance | Daily assessments from baseline up to day 7
  Mean days to pain disappearance in the treatment group respect to placebo
Pain free patients percentage | Daily assessments from baseline up to day 7
  Percentage of patients who will report to be pain free according to the VAS scale
Ulcers reduction | Daily assessments from baseline up to day 7
  Reduction of the number of ulcers respect to baseline
Lesions healing percentage | Daily assessments from baseline up to day 7
  Percent of lesions with complete healing
Pain reduction | From baseline up to day 7
  Reduction of pain (immediate relief on application, no burning sensation, measurement of how many days pain persists)
Safety | From baseline up to day 7
  Number of Adverse Events and Serious Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico "Umberto I" - U.O.C. di Odontoiatria Pediatrica ed Odontostomatologia, Rome, Italy